CLINICAL TRIAL: NCT05952440
Title: Dissecting the Cellular and Molecular Atlas of Rheumatoid Arthritis in Sustained Remission to Identify Pathways Maintaining Remission and Triggering Flares
Acronym: FLARE-RA
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: University of Glasgow (Other); Fundacion Clinic per a la Recerca Biomédica (Other); Newcastle University (Other)
Responsible Party: Sponsor
Other Study IDs: 5600
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- RA in remission who performed synovial biopsy before treatment change
  Interventions: Other: Tapering and/or discontinuation of treatment based on standard of care; Other: No tapering and/or discontinuation of treatment based on standard of care
- RA in remission eligible to synovial biopsy before treatment change
  Interventions: Other: Tapering and/or discontinuation of treatment based on AI-guidance; Other: No tapering and/or discontinuation of treatment based on AI-guidance; Other: Tapering and/or discontinuation of treatment based on standard of care; Other: No tapering and/or discontinuation of treatment based on standard of care
- Subjects asymptomatic for joint inflammation without ACPA/RF positivity

INTERVENTIONS:
Other: Tapering and/or discontinuation of treatment based on AI-guidance — After synovial tissue biopsy, pharmacological treatment (cDMARDs or bDMARDs) are tapered first and then bDMARDs and/or cDMARDs are discontinued based on AI-guidance
  Groups: RA in remission eligible to synovial biopsy before treatment change
Other: No tapering and/or discontinuation of treatment based on AI-guidance — Ongoing therapeutic are not changed (tapered or discontinued) after synovial biopsy performance based on AI-guidance
  Groups: RA in remission eligible to synovial biopsy before treatment change
Other: Tapering and/or discontinuation of treatment based on standard of care — After synovial tissue biopsy, pharmacological treatment (cDMARDs or bDMARDs) are tapered first and then bDMARDs and/or cDMARDs are discontinued based on standard of care
  Groups: RA in remission eligible to synovial biopsy before treatment change; RA in remission who performed synovial biopsy before treatment change
Other: No tapering and/or discontinuation of treatment based on standard of care — Ongoing therapeutic are not changed (tapered or discontinued) after synovial biopsy performance based on standard of care
  Groups: RA in remission eligible to synovial biopsy before treatment change; RA in remission who performed synovial biopsy before treatment change

SUMMARY:
The FLARE-RA study will have the following research objectives:

A) To establish the cellular and molecular atlas of remission RA achieved with different therapeutics aimed to identify (i) cell clusters/pathways driving disease flare or maintaining remission and (ii) provide an evidence base for developing ML tools for predicting flares.

B) To test the performance of a ML-derived algorithm on longitudinal remission RA cohort in a biopsy-driven study.

C) To dissect the cellular and molecular mechanisms of remission maintenance and joint flares.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid Arthritis classified based on the 2010 EULAR/ACR Classification Criteria
* Stable treatment with cDMARDs and/or bDMARDs (≥12 months)
* Stable remission status (at least DAS28-CRP<2.6) (≥6 months)
* No concomitant steroid treatment (≥6 months)
* Absence of Power-Doppler signal at ultrasound assessment (wrist, MCP, PIP, Knee, ankle and II-V MTP bilaterally) in 3 evaluations 3 months apart.

Exclusion Criteria:

* DAS28-CRP≥2.6
* Presence of Power-Doppler signal ≥1 at ultrasound assessment (wrist, MCP, PIP, Knee, ankle and II-V MTP bilaterally)
* Other chronic inflammatory disease

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Experimental groups will include, the following classes of patients:
  1. Rheumatoid Arthritis in sustained clinical and ultrasound remission afferent to the Division of Rheumatology - Fondazione Policlinico Universitario A. Gemelli IRCCS, in Rome who already underwent synovial tissue biopsy for the routine clinical assessment of tissue inflammation (retrospective cohort) (n=40).
  2. Rheumatoid Arthritis in sustained clinical and ultrasound remission afferent to the Division of Rheumatology - Fondazione Policlinico Universitario A. Gemelli IRCCS, in Rome or to the Hospital Clinic and Fundació Clinic per la Recerca Biomèdica, in Barcelona eligible to synovial tissue biopsy for the routine clinical assessment of tissue inflammation (prospective cohort) (n=40 for each center).
  3. Subjects asymptomatic for joint inflammation without ACPA/RF positivity (n=10) (University of Glasgow).
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2026-05-10 (Estimated); Study Completion 2026-05-10 (Estimated)

PRIMARY OUTCOMES:
Establishment of cellular and molecular atlas of remission RA | months 1-12
  To establish the cellular and molecular atlas of remission RA achieved with different therapeutics aimed to identify (i) cell clusters/pathways driving disease flare or maintaining remission and (ii) provide an evidence base for developing ML tools for predicting flares.

SECONDARY OUTCOMES:
To test the performance of a ML-derived algorithm on longitudinal remission RA cohort in a biopsy-driven study. | months 13-36
  To test the performance of a ML-derived algorithm on longitudinal remission RA cohort in a biopsy-driven study.
To dissect the cellular and molecular mechanisms of remission maintenance and joint flares | months 13-36
  To dissect the cellular and molecular mechanisms of remission maintenance and joint flares in in vivo and in vitro systems

CONTACTS AND LOCATIONS:
Locations (4):
- Division of Rheumatology, Rome, Italy
- Hospital Clinic and Fundació Clinic per la Recerca Biomèdica, Barcelona, Spain
- United Kingdom (2):
  - Research into Inflammatory Arthritis Centre Versus Arthritis (RACE), Glasgow
  - Newcastle University, Newcastle upon Tyne